CLINICAL TRIAL: NCT05186077
Title: Brain Circuitry Analysis in Bipolar Disorder
Status: Terminated | Type: Observational
Why Stopped: The original funding for this study ended and we were not able to secure new funding to continue
Sponsor: Jennifer Sweet (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jennifer Sweet, Principal Investigator, Case Western Reserve University
Organization: Case Western Reserve University (Other)
Other Study IDs: STUDY20201112; 1R56MH121598-01A1 (NIH)
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Controls: These participants will not have any psychiatric disorder as assessed by a structured clinical interview for psychiatric disorders.
  Interventions: Other: Magnetic Resonance Imaging
- Treatment-Responsive BD: This group will be composed of participants who have BDI or BDII and have most recently been depressed but are currently in remission with evidence-based treatments for bipolar disorder
  Interventions: Other: Magnetic Resonance Imaging; Other: Psychiatric testing; Other: Eye-Tracking; Other: Neuropsychology Evaluation
- Treatment-Refractory BD: This group will be composed of participants who have BDI or BDII, are currently depressed or manic with their current episode lasting at least 6months and not responding to 2 or more adequate evidence-based treatments for BDI or BDII.
  Interventions: Other: Magnetic Resonance Imaging; Other: Psychiatric testing; Other: Eye-Tracking; Other: Neuropsychology Evaluation

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Imaging data for research purposes (high-resolution T1 structural and DWI MRI) will be acquired
Other: Psychiatric testing — Subjects will be evaluated using psychiatric assessments
  Groups: Treatment-Refractory BD; Treatment-Responsive BD
Other: Eye-Tracking — Eye-tracking assessments will be done to biases toward positive and negative stimuli including images of neutral, fearful/threatening, sad, and happy.
  Groups: Treatment-Refractory BD; Treatment-Responsive BD
Other: Neuropsychology Evaluation — The neuropsychology evaluation will measure verbal learning/memory, attention/working memory, psychomotor speed, verbal fluency/processing speed, and executive function
  Groups: Treatment-Refractory BD; Treatment-Responsive BD

SUMMARY:
The goal of this cross-sectional study is to use diffusion-weighted imaging based tractography (DWT) to assess white matter (WM) pathways in treatment-refractory bipolar disorder (REF-BD) and treatment responsive bipolar disorder (RSP-BD) subjects compared to healthy controls (HCs). This project will include a prospective controlled trial to include 50 subjects with REF-BD, 50 patients RSP-BD and 50 healthy volunteers.

ELIGIBILITY:
Group 1: Healthy Volunteers

Inclusion Criteria for Group 1:

1. Male or female ≥18 years of age
2. Capable of understanding/complying with protocol requirements
3. Has competency to understand and sign informed consent form
4. Physically healthy with no acute medical condition and ≤3 stable, chronic medical conditions
5. Without current and/or lifetime psychiatric disorders as assessed by the Mini International Neuropsychiatric Interview for DSM-5 (MINI)

Exclusion Criteria for Group 1:

1. Acute medical condition or >3 stable, chronic health conditions
2. Significant structural brain lesion
3. Progressive neurological disease
4. Preexisting implanted electrical device
5. Currently pregnant or planning to become pregnant
6. Contraindications to MR imaging
7. Tests positive for cannabis, illegal substances, or prescription medications without valid prescription
8. Currently taking steroids, opioids, or other agents that might affect brain circuitry per research team discretion
9. Use of cigarettes or other nicotine products within 12 hours of imaging visit
10. Use of stimulants 24 hours prior MRI visit
11. Presents an immediate danger to self or others as judged by research psychiatrist
12. Has psychiatric disorder, including alcohol/drug use disorder or personality disorder

Group 2: Treatment-Responsive BDI

Inclusion Criteria for Group 2:

1. Male or female ≥18 years of age
2. Capable of understanding/complying with protocol requirements
3. Has competency to understand and sign informed consent form
4. Physically healthy with no acute medical condition and ≤3 stable, chronic medical conditions
5. Meets diagnostic criteria for BDI or BDII according to the DSM-5 criteria
6. Must be stable on current BD medications with no dosing changes in the last 30 days or not currently taking any BD medications.
7. Recent mood episode must currently be in remission for > 8 weeks
8. Montgomery-Asberg Depression Rating Scale (MADRS) ≤10 total score during the psychiatric assessments portion and at the MRI visit (if repeated at MRI visit)
9. Young Mania Rating Scale (YMRS) ≤12 total score during the psychiatric assessments portion and at the MRI visit (if repeated at MRI visit)
10. Clinical Global Impression-Severity for Bipolar Disorder (CGI-S-BD) ≤2 during the psychiatric assessments visit
11. Must be adherent (≥ 80%) with BD medication(s)

Exclusion Criteria for Group 2:

1. Acute medical condition or >3 stable, chronic health conditions
2. Significant structural brain lesion
3. Progressive neurological disease
4. Preexisting implanted electrical device
5. Currently pregnant or planning to become pregnant
6. Contraindications to MR imaging
7. Tests positive for cannabis, illegal substances, or prescription medications without valid prescription
8. Currently taking steroids, opioids, or other agents that might affect brain circuitry per research team discretion
9. Use of cigarettes or other nicotine products within 12 hours of imaging visit
10. Use of stimulants within 24 hours of imaging visit
11. Presents an immediate danger to self or others as judged by research psychiatrist
12. Has had changes in medications within 30 days
13. Contribution of any co-occurring psychiatric comorbidity disproportionate to contribution of BDI or BDII
14. Meets DSM-5 criteria for current borderline or antisocial personality disorder
15. Meets DSM-5 criteria for alcohol and/or drug use disorder within 6 months, excluding caffeine and/or nicotine

Group 3: Treatment-Refractory BDI

Inclusion Criteria for Group 3:

1. Male or female ≥18 years of age
2. Capable of understanding/complying with protocol requirements
3. Has competency to understand and sign informed consent form
4. Physically healthy with no acute medical condition and ≤3 stable, chronic medical conditions
5. Meets diagnostic criteria for BDI or BDII according to the DSM-5 criteria
6. Must be stable on drugs, including at least 1 mood stabilizer, with no dosing changes in the last 30 days
7. GCI-S-BD >3 at the psychiatric assessments visit
8. MADRS ≥20 total score or YMRS ≥18 total score during the psychiatric assessments portion and at the MRI visit (if repeated at MRI visit)
9. BD-associated mood episodes are primary source of disability, according to both subject and psychiatrist
10. Current depressive episode lasting ≥6 months despite ≥ 2 adequate evidence-based first-line treatment > 8 weeks, current manic/hypomanic episode lasting ≥2 months despite ≥ 2 adequate evidence-based first-line treatment > 4 weeks, or meeting rapid cycling criteria in last 12 months despite ≥2 evidence-based first-line treatments for BDI or BDII assessed with assistance of Modified Antidepressant Treatment History Form (MATHF)
11. Severe impairment with score of ≥7 on at least one of three subscales of Sheehan Disability Scale (SDS), which includes assessment of work-life, family-life, and social life during the psychiatric assessments portion

Exclusion Criteria for Group 3:

1. Acute medical condition or >3 stable, chronic health conditions
2. Significant structural brain lesion
3. Progressive neurological disease
4. Preexisting implanted electrical device
5. Currently pregnant or planning to become pregnant
6. Contraindications to MR imaging
7. Tests positive for cannabis, illegal substances, or prescription medications without valid prescription
8. Currently taking steroids, opioids, or other agents that might affect brain circuitry per research team discretion
9. Use of cigarettes or other nicotine products within 12 hours of imaging visit
10. Use of stimulants within 24 hours of imaging visit
11. Presents an immediate danger to self or others as judged by research psychiatrist
12. Has had changes in medications within 30 days
13. Contribution of any co-occurring psychiatric comorbidity disproportionate to contribution of BDI or BDII
14. Meets DSM-5 criteria for current borderline or antisocial personality disorder
15. Meets DSM-5 criteria for alcohol and/or drug use disorder within 6 months, excluding caffeine and/or nicotine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from all three groups will be made up of those who respond to IRB approved advertisements or are referred by a provider within the UHCMC Department of Psychiatry or other provider referral.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Characterize white matter (WM) connectivity with DWT to identify an anatomical substrate for BD that has future potential as a therapeutic target | Day 1
  The imaging visit will consist of an MRI with diffusion-weighted imaging (DWI) sequences

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sweet, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States